CLINICAL TRIAL: NCT02597361
Title: Angiotensin II Receptor Blockade in Vascular Ehlers Danlos Syndrome: a Double Blind, Randomized, Placebo Controlled, Multicenter Trial.
Brief Title: Angiotensin II Receptor Blockade in Vascular Ehlers Danlos Syndrome (ARCADE)
Acronym: ARCADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P140918; 2015-001065-76 (EudraCT Number)
Record Dates: First submitted 2015-10-23; First posted 2015-11-05 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2020-10

CONDITIONS: Ehlers-Danlos Syndrome, Vascular Type
Keywords: Ehlers-Danlos syndrome, vascular type; Type 2 Angiotensin Receptor Blockers
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irbesartan (Active Comparator): Irbesartan: 150 or 300 mg o.d. for 2 years.The up-titration of irbesartan from 150 mg to 300 mg o.d. occurs during the first 8 weeks following randomization and will be driven by clinical, hemodynamic and biological (plasma creatinine and K) tolerability.
  Interventions: Drug: Irbesartan
- Placebo (Placebo Comparator): Placebo once or twice per day for 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irbesartan — Irbesartan: 150 or 300 mg o.d. The up-titration of irbesartan from 150 mg to 300 mg o.d. occur during the first 8 weeks following randomization
  Arms: Irbesartan
Drug: Placebo — Placebo o.d. to match 150mg or 300mg irbesartan tablets
  Arms: Placebo

SUMMARY:
This study aims to verify the hypothesis that patients with Vascular Ehlers Danlos syndrome (vEDS) should benefit of the blockade of angiotensin (Ang) II noxious effects on their vasculature affected by a defect in type III collagen in addition to the effects celiprolol. This randomized, double blind, placebo controlled trial compares the administration of the Ang II type I receptor blocker (ARB) - irbesartan- to placebo over a 2-year period in vEDS patients with the main objective to reduce the incidence of both symptomatic and asymptomatic vascular events.

DETAILED DESCRIPTION:
vEDS is a rare life-threatening inherited condition due to mutations at the COL3A1 gene encoding the pro-alpha 1 chain of type III procollagen (OMIM #130050) with unpredictable and recurring arterial dissections/aneurysms starting in the early adulthood. The investigators have previously shown that a treatment with 200-400 mg per day of celiprolol, reduces both fatal and non-fatal vascular events in patients with vEDS. If tolerated, the treatment is now the standard treatment for vEDS. However, despite celiprolol , symptomatic and asymptomatic arterial events continue to occur in vEDS patients. Recent findings suggest a possible deleterious effect of endogenous Angiotensin II on medium size arteries in vEDS patients. The hypothesis of this study is that the blockade of endogenous Ang II will provide supplemental vascular protection and thus reduce recurrence of arterial events in vEDS patients.

The primary objective of this study is to determine in patients with molecularly proven vEDS, whether an Ang II receptor blocker, prescribed at an optimally tolerated dose combined with the reference celiprolol treatment, decreases the 24 months rate of both asymptomatic and symptomatic cardiovascular (CV) events when compared to placebo.

Methodology:

Multicenter, double-blind, randomized (1:1), placebo-controlled, parallel group, study with blind endpoint evaluation in adult vEDS patients.

Main criteria for inclusion:

Patients of both sexes aged 18 to 70 years with molecularly proven vEDS, not in an acute phase of the disease, with no contra-indication for taking an Ang II blocker.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically-proven vEDS (presence of a pathogenic mutation at the COL3A1 gene);
* Age ≥18 years and <70 years;
* Men and women with reliable contraception or negative beta-HCG at screening;
* Celiprolol at the optimal tolerated dose since at least 12 weeks;
* vEDS patient fully intolerant to celiprolol but not treated with any other drug active on the vascular system, except another beta-blocker;
* No compelling indication for ARB therapy (renal infarction, hypertension, proteinuric nephropathy, chronic heart failure, myocardial infarction, stroke);
* Estimated glomerular filtration rate (GFR) ≥ 30ml/min/1,73m2 (MDRD Formula);
* Normal or clinically acceptable 12-lead ECG;
* Written informed consent to participate in the study.

Exclusion Criteria:

General criteria

* Unlikely to co-operate in the study and/or poor compliance anticipated by the investigator, e.g., uncooperative attitude, inability to return for follow-up visit, and unlikelihood of completing the study;
* Participation in another interventional therapeutic study at the same time or within 3 months prior to the beginning of the present study;
* Participant not affiliated to the French social security;
* No written informed consent;
* Severe contrast media allergy, not amenable to pre-treatment Medical and therapeutic criteria
* History of previous symptomatic visceral complication (any CV event, pulmonary or digestive event) in the 3 months preceding the inclusion;
* Formal indication for an antihypertensive medication (office BP ≥140/90 mmHg on celiprolol on at least two separated visits, confirmed by daytime ambulatory BP or home BP ≥ 135/85 mmHg);
* Concomitant treatment with renin-angiotensin-aldosterone system blocking agents apart from the study drug, e.g. ACEI, ARB or aldosterone-antagonist or any renin inhibitor, if given for an elective indication (heart failure, renal infarction, chronic kidney disease, proteinuria, myocardial infarction, stroke);
* Any cardiac condition that justifies a specific medical care (i.e. second or third degree auriculo-ventricular block, potentially life threatening arrhythmia or other uncontrolled arrhythmia or persistent arrhythmia, clinically significant valvular heart disease);
* Known significant renal artery stenosis with evidence of renal ischemia (on Duplex ultrasound, CTA, or other exam);
* Any concurrent life threatening condition other than vEDS with a life expectancy less than 2 years;
* Likely allergy or hypersensitivity to irbesartan, based on known allergies to drugs of the same class, or which in the opinion of the investigator suggests an increased potential for an adverse hypersensitivity as well as known or suspected contraindications to the study drug;
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety;
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human Chorionic Gonadotropin (hCG) laboratory test (>5 mIU/ml);
* Women of child-bearing potential (WOCBP) without reliable contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Cardiovascular morbidity and mortality | 2 years
  Total number of any non-fatal and fatal cardiovascular events or events related to vEDS
Arterial lesions | 2 years
  number and severity of arterial lesions detected by CTA

SECONDARY OUTCOMES:
Rate of any symptomatic cardiovascular event | 2 years
  CV death; any morbid and fatal events related to vEDS; Any non fatal CV event; Non-fatal stroke
Occurrence of new asymptomatic arterial lesions (aneurysm, dissection), detected by a systematic CTA | 2 years
  Arterial dissection/rupture/aneurysm in any vascular bed
Time to first symptomatic clinical morbid and fatal events | 2 years
Number of unplanned hospitalization for any vEDS related event | 2 years
Total number of arterial lesions detected by vascular DUS | 2 years
  Echo duplex ultrasound made at inclusion, 6, 12, 18 and 24 months
Total number of arterial lesions worsened during follow-up | 2 years
Changes in PWV (Pulse Wave Velocity) | 2 years
  Applanation tonometry made at randomization visit, 6, 12, 18 and 24 months
Changes in large arteries properties (diameter, wall stress, stiffness) | 2 years
  Echotracking made at randomization visit, 6, 12, 18 and 24 months
Decrease in office systolic/diastolic BP | 2 years
  Vital signs (BP and HR) measured by automatic device at each visit
Change in estimated glomerular filtration rate (MDRD) | 2 years
  eGFR evaluated at each visit
Tolerability and safety of the irbesartan assessed by orthostatic hypotension, plasma creatinine, plasma K+ evaluated at each visit | 2 years
Compliance to treatment | 2 years
  Spot urine for drug determination (celiprolol and irbesartan urinary detection) made at randomization visit and 3, 12 and 24 months
Quality of life | 2 years
  SF36 and HADS questionnaires submitted to participants at randomization visit, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier JEUNEMAITRE, MD,PHD, Principal Investigator — AP-HP, INSERM
Locations (15):
- France (15):
  - CHU DE BORDEAUX - Hopital Saint Andre, Bordeaux
  - CHU DE LYON - Hopital Femme Mere Enfant, Bron
  - CHU DE CAEN - Hopital Cote de Nacre, Caen
  - CHU DE TOURS - Hopital Trousseau, Chambray-lès-Tours
  - CHU DE GRENOBLE - Hopital Albert Michallon, Grenoble
  - CHU DE GRENOBLE - Hopital Couple Enfant, Grenoble
  - CHRU DE LILLE - Hopital Claude Huriez, Lille
  - CHU DE LYON - Hopital Edouard Herriot, Lyon
  - AP-HM - Hopital de la Timone, Marseille
  - CHU DE MONTPELLIER - Hopital Saint Eloi, Montpellier
  - CHU DE NANTES - Hopital Hotel-Dieu, Nantes
  - AP-HP - Hopital Europeen Georges-Pompidou, Paris
  - CHU DE TOULOUSE - Hopital Purpan, Toulouse
  - CHU DE TOULOUSE - Hopital Rangueil, Toulouse
  - CHRU DE NANCY - Institut Lorrain du Coeur et des Vaisseaux, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results reported in publications after de-identification (text, tables, figures, and appendices).
  IPD detailed in the protocol of a planned meta-analysis could be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years following publication. No end date
Access Criteria: With whom? Qualified researchers who provide a methodologically sound proposal. Collaboration with the original team will be fostered.
  For what types of analyses? To achieve aims in the approved proposal. Meta-analyses are encouraged.
  By what mechanism will data be made available? Data sharing must be accepted by the sponsor and the principal investigator (PI) based on scientific project and scientific involvement of the PI team. Proposals should be directed to xavier.jeunemaitre@aphp.fr. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory data access agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Frank M, Albuisson J, Ranque B, Golmard L, Mazzella JM, Bal-Theoleyre L, Fauret AL, Mirault T, Denarie N, Mousseaux E, Boutouyrie P, Fiessinger JN, Emmerich J, Messas E, Jeunemaitre X. The type of variants at the COL3A1 gene associates with the phenotype and severity of vascular Ehlers-Danlos syndrome. Eur J Hum Genet. 2015 Dec;23(12):1657-64. doi: 10.1038/ejhg.2015.32. Epub 2015 Mar 11. PMID 25758994
- [Result] Faugeroux J, Nematalla H, Li W, Clement M, Robidel E, Frank M, Curis E, Ait-Oufella H, Caligiuri G, Nicoletti A, Hagege A, Messas E, Bruneval P, Jeunemaitre X, Bergaya S. Angiotensin II promotes thoracic aortic dissections and ruptures in Col3a1 haploinsufficient mice. Hypertension. 2013 Jul;62(1):203-8. doi: 10.1161/HYPERTENSIONAHA.111.00974. Epub 2013 Apr 29. PMID 23630948
- [Result] Ong KT, Perdu J, De Backer J, Bozec E, Collignon P, Emmerich J, Fauret AL, Fiessinger JN, Germain DP, Georgesco G, Hulot JS, De Paepe A, Plauchu H, Jeunemaitre X, Laurent S, Boutouyrie P. Effect of celiprolol on prevention of cardiovascular events in vascular Ehlers-Danlos syndrome: a prospective randomised, open, blinded-endpoints trial. Lancet. 2010 Oct 30;376(9751):1476-84. doi: 10.1016/S0140-6736(10)60960-9. Epub 2010 Sep 7. PMID 20825986
- [Derived] Jeunemaitre X, Mousseaux E, Frank M, Adham S, Pitocco F, Billon C, Ben Yakhlef M, El Hachmi M, Bura-Riviere A, Lapebie FX, Le Hello C, Laneelle D, Seinturier C, Dieterich K, Lambert M, Dupuis-Girod S, Zuily S, Bal-Theoleyre L, Boulon C, Henneton P, Lu E, Denarie N, Boutouyrie P, Mirault T, Chatellier G, Azizi M. Efficacy of Irbesartan in Celiprolol-Treated Patients With Vascular Ehlers-Danlos Syndrome. Circulation. 2025 Mar 11;151(10):686-695. doi: 10.1161/CIRCULATIONAHA.124.072849. Epub 2025 Feb 5. PMID 39906986